CLINICAL TRIAL: NCT06012799
Title: Prospective Observational Study for Efficacy of Perioperative Serum Glucose Level Evaluated by Continuous Glucose Monitoring System in Kidney Transplantation Patients
Brief Title: Continuous Glucose Monitoring in Peri-operative Period in Kidney Transplant Recipients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SNUH-CGM-KT-V1.2
Record Dates: First submitted 2023-08-22; First posted 2023-08-25 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-08

CONDITIONS: New Onset Diabetes After Transplantation
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Diagnostic Test: continuous glucose monitoring — FreeStyle Libre Flash Glucose Monitoring System

SUMMARY:
his study aims to utilize Continuous Glucose Monitoring (CGM) to observe glucose fluctuations in kidney transplant recipients and predict New-Onset Diabetes After Transplantation (NODAT) based on these patterns. Additionally, it seeks to investigate glucose variability resulting from medications and surgeries such as immunosuppressants and steroid regimens post-kidney transplantation. This prospective observational study anticipates identifying factors influencing blood glucose levels and contributing to future research on blood glucose management using CGM monitoring in kidney transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* The study will target 100 kidney transplant patients who have provided consent, among those who underwent the procedure at Seoul National University Hospital after March 2021.

Exclusion Criteria:

* multi-organ transplant
* history of previous kidney transplant
* less than 18 years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Kidney transplant patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of NODAT | 6 months after kidney transplantation
  rate of new onset diabetes after transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No